CLINICAL TRIAL: NCT04579783
Title: Comparison of Corticosteroid and Repeated Dextrose Hydro-dissection for Carpal Tunnel Syndrome Patients
Brief Title: Corticosteroid and Repeated Dextrose Hydro-dissection for Carpal Tunnel Syndrome Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 202007021MINB
Record Dates: First submitted 2020-09-27; First posted 2020-10-08 (Actual); Last update posted 2021-12-15 (Actual); Status verified 2021-12

CONDITIONS: Carpal Tunnel Syndrome
Keywords: Hydro-dissection; Dextrose; Corticosteroid
MeSH Terms: conditions — Carpal Tunnel Syndrome | interventions — Triamcinolone Acetonide; Glucose; Water

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ultrasound intracarpal corticosteroid injection (Active Comparator): Twice ultrasound-guided hydro-dissection of median nerve at carpal tunnel level.
  1st injection (0 week): 40mg triamcinolone acetonide (40mg/mL ) with 4mL normal saline, 2nd injection (6 week): 5 mL normal saline
  Interventions: Drug: Triamcinolone Acetonide
- Ultrasound guided intracarpal dextrose hydro-dissection (Active Comparator): Twice ultrasound-guided hydro-dissection of median nerve at carpal tunnel level.
  Group B: 1st injection (0 week): 5 mL 5% dextrose, 2nd injection (6 week): 5 mL 5% dextrose
  Interventions: Drug: Dextrose 5% in water

INTERVENTIONS:
Drug: Triamcinolone Acetonide — Group A: 40mg triamcinolone acetonide (1mL) + 4mL normal saline
  Other Names: Shincort
  Arms: Ultrasound intracarpal corticosteroid injection
Drug: Dextrose 5% in water — Group B: 5mL 5% dextrose
  Other Names: Vitagen
  Arms: Ultrasound guided intracarpal dextrose hydro-dissection

SUMMARY:
Carpal tunnel syndrome (CTS) is the most prevalent peripheral nerve entrapment of upper limb. Typical symptoms comprise pain, numbness or tingling of the thumb and index, middle or ring fingers. Thumb weakness and decreased grip strength can occur in the later stage. Currently treatments included physical modalities (low power laser, transcutaneous electrical nerve stimulation, ultrasound), medication, splinting, injection and surgery. Ultrasound guided intracarpal hydro-dissection of median nerve had been proposed based on its accurate localization, while the injectates were diverse. Corticosteroid has been widely used for CTS for decades. However, growing evidences suggested that 5% dextrose, normal saline, platelet rich plasma injection also have therapeutic effects on alleviating CTS symptoms. Among the injectates, a single 5% dextrose injection could be considered as a substitute of corticosteroid based on its long term effect up to six months. However, the clinical efficacy of 5% dextrose injection has not validated by the further study. The investigators aim to compare the therapeutic effect of 5% dextrose injection with corticosteroid injection in patients with CTS, up to 12 weeks follow up.

DETAILED DESCRIPTION:
Introduction:

Carpal tunnel syndrome (CTS) is the most prevalent peripheral nerve entrapment of upper limb. Typical symptoms comprise pain, numbness or tingling of the thumb and index, middle or ring fingers. Thumb weakness and decreased grip strength can occur in the later stage. Currently treatments included physical modalities (low power laser, transcutaneous electrical nerve stimulation, ultrasound), medication, splinting, injection and surgery. Ultrasound guided intracarpal hydro-dissection of median nerve had been proposed based on its accurate localization, while the injectates were diverse. Corticosteroid has been widely used for CTS for decades. However, growing evidences suggested that 5% dextrose, normal saline, platelet rich plasma injection also have therapeutic effects on alleviating CTS symptoms. Among the injectates, a single 5% dextrose injection could be considered as a substitute of corticosteroid based on its long term effect up to six months. However, the clinical efficacy of 5% dextrose injection has not validated by the further study. Whether repeated injection could expand the treatment effect was undetermined. The investigators aim to compare the therapeutic effect repeated 5% dextrose injection with corticosteroid injection in patients with CTS, up to 12 weeks follow up.

Material and methods:

Participants: 60 adult patients (>20 year olds) with carpal tunnel syndrome, recruited from outpatient clinic.

Inclusion criteria: Presenting with CTS symptoms, including nocturnal, postural, or motion-associated paresthesias +/- pain of the median nerve distribution area in the subjective hand. Confirmed Electrophysiological confirmed median neuropathy at the wrist with mild to moderate degree. Persistent symptoms for more than 3 months

Exclusion Criteria: Patients cervical radiculopathy, polyneuropathy, brachial plexopathy, thoracic outlet syndrome. Recent corticosteroid injection to the carpal tunnel within 6 months.

Thenar muscle atrophy. Previous history of carpal tunnel surgical release. History of wrist trauma. Regular use of systemic nonsteroidal anti-inflammatory drugs, corticosteroids or diuretics. Pregnancy. Cognitive impairment.

Objective:

The aim of this study is to compare the treatment effect of repeated 5 mL 5% dextrose with 5mL triamcinolone acetonide injection in patients with CTS.

Detail of the intervention The study is designated as randomized, double blinded, and parallel experiment. The randomization was decided by random table in block of 4.

Repeated ultrasound guided injection intracarpal median nerve hydro-dissection with 5 mL 5% dextrose (Group B) or 5mL triamcinolone acetonide injection (Group A) in patients with CTS.

The regimen was shown as below:

Group A: 1st injection (0 week): 40mg triamcinolone acetonide (40mg/mL) with 4mL normal saline, 2nd injection (6 week): 5 mL normal saline Group B: 1st injection (0 week): 5 mL 5% dextrose, 2nd injection (6 week): 5 mL 5% dextrose

Skin infiltration with local anesthetic (lidocaine cream) at the needle insertion site was performed before the injection. Then injection was performed after sterilization. The equipment for ultrasound-guided injection will be high-resolution ultrasound machine with the linear probe.

Outcome measurement:

Boston Carpal Tunnel Syndrome Questionnaire (BCTQ) and Visual analogue scale (VAS) before 1st injection, before 2nd injection (6-week) and 12-week after first injection.

Electrophysiological evaluation (amplitude and distal latency of median nerve compound motor action potential and sensory nerve action potential); cross-sectional area of median nerve at carpal tunnel inlet, were evaluated before and 12-week after 1st injection.

Global assessment of treatment was evaluated at before 2nd injection (6-week) and 12-week after first injection.

Statistical analysis:

Continuous variables Student's t test: fit assumption of normal distribution Mann-Whitney test: does not fit the assumption of normal distribution Categorical variables (1) Chi-square test (2) Fisher exact test: sparse data (3)Repeated-measures analysis of variance (ANOVA) was used to evaluate the effect of injection with post-hoc Bonferroni test to evaluate intra-group data at different time-frame

Keywords: Hydro-dissection, corticosteroid, dextrose, carpal tunnel syndrome

ELIGIBILITY:
Inclusion Criteria:

* Presenting with carpal tunnel syndrome symptoms, including nocturnal, postural, or motion-associated paresthesias +/- pain of the median nerve distribution area in the subjective hand
* Confirmed Electrophysiological confirmed median neuropathy at the wrist with mild to moderate degree
* Persistent symptoms for more than 3 months

Exclusion Criteria:

* Patients with suspicious of CTS mimic condition, including cervical radiculopathy, polyneuropathy, brachial plexopathy, thoracic outlet syndrome
* Recent corticosteroid injection to the carpal tunnel within 6 months
* Thenar muscle atrophy
* Previous history of carpal tunnel surgical release
* History of wrist trauma
* Regular use of systemic nonsteroidal anti-inflammatory drugs, corticosteroids or diuretics
* Pregnancy
* Cognitive impairment

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-11-27 (Actual); Primary Completion 2022-10 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Boston Carpal Tunnel Syndrome Questionnaire | Change of the score between 6 weeks and baseline(1st injection), and change of the score between 12 weeks and baseline (1st injection))
  Evaluation of symptom severity (11-question) and functional impairment (8-question) subscale. The scores range from 0 to 5 points for each question, with higher scores indicating greater severity and dysfunction.

SECONDARY OUTCOMES:
Visual analogue scale | Change of the score between 6 weeks and baseline(1st injection), and change of the score between 12 weeks and baseline (1st injection))
  Pain intensity evaluation, from 0 to 10 points, a 11-point scale. The higher scores indicate severe pain.
Distal latency of median nerve sensory nerve action potential (Unit: ms) | change of the score between 12 weeks and baseline (1st injection)
  recoding at index finger by antidromic stimulation
Amplitude of median nerve sensory nerve action potential (Unit: μV) | change of the score between 12 weeks and baseline (1st injection)
  recording at index finger by antidromic stimulation
Distal latency of median nerve compound motor action potential (Unit: ms) | change of the score between 12 weeks and baseline (1st injection)
  recording at abductor pollicis brevis muscle
Amplitude of median nerve compound motor action potential (Unit: mV) | change of the score between 12 weeks and baseline (1st injection)
  recording at abductor pollicis brevis muscle
Cross-sectional area of median nerve (unit: mm2) | Change of the score between 6 weeks and baseline(1st injection), and change of the score between 12 weeks and baseline (1st injection))
  Ultrasound evaluation of the median nerve size
Global assessment of treatment (1st) | 6-week after 1st injection (before 2nd injection)
  self-reported global assessment of treatment on 5 category (much improved, improved, no change, worse, or much worse)
Global assessment of treatment (2nd) | 6-week after 2nd injection (12-week after 1st injection)
  self-reported global assessment of treatment on 5 category (much improved, improved, no change, worse, or much worse)

CONTACTS AND LOCATIONS:
Overall Officials: Ke-Vin Chang, MD,PhD, Principal Investigator — National Taiwan University Hospital Beihu Branch
Locations (1):
- National Taiwan University Hospital, Bei-Hu Branch, Taipei, Wanhua District, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wu YT, Ho TY, Chou YC, Ke MJ, Li TY, Tsai CK, Chen LC. Six-month Efficacy of Perineural Dextrose for Carpal Tunnel Syndrome: A Prospective, Randomized, Double-Blind, Controlled Trial. Mayo Clin Proc. 2017 Aug;92(8):1179-1189. doi: 10.1016/j.mayocp.2017.05.025. PMID 28778254